CLINICAL TRIAL: NCT07123090
Title: A Phase 2 Study of Sasanlimab, Palbociclib and Axitinib in Metastatic Renal Cell Carcinoma - SPARCC
Brief Title: A Phase 2 Study of Sasanlimab, Palbociclib and Axitinib in Metastatic Renal Cell Carcinoma
Acronym: SPARCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie Berg (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Stephanie Berg, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-258
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Renal Cancer; Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer; Translocation Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; Metastatic Renal Cancer; Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer; Translocation Renal Cell Carcinoma; ccRCC; tRCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — palbociclib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sasanlimab, Axitinib, and Palbociclib (Experimental): A Bayesian dose-limiting toxicity plan will be employed per protocol with a monitoring time period of the first two cycles of therapy and starting after the first three participants have started protocol therapy. 25 enrolled participants will complete:
  * Baseline visit with assessments and imaging
  * Imaging every 8 weeks for 16 weeks, then every 12 weeks
  * Cycle 1 Through End of Treatment (28 day cycles):
    * Day 1: Predetermined dose of Sasanlimab 1x daily
    * Days 1 through 28: Predetermined dose of Axitinib 2x daily,
    * Days 8 through 28: Predetermined dose of Palbociclib 1x daily
  * End of treatment visit
  * Follow up every 6 months for 2 years after treatment discontinuation
  Interventions: Drug: Sasanlimab; Drug: Palbociclib; Drug: Axitinib

INTERVENTIONS:
Drug: Sasanlimab — Recombinant humanized monoclonal antibody, prefilled syringe, subcutaneous (under the skin) injection per protocol
  Other Names: PF-06801591
Drug: Palbociclib — Cyclin-dependent kinase (CDK) 4/6 inhibitor, tablet taken orally per protocol
  Other Names: C24H29N7O2
Drug: Axitinib — Vascular endothelial growth factor (VEGF) inhibitor, tablet taken orally per standard of care
  Other Names: C22H18N4OS

SUMMARY:
The goal of this research study is to evaluate how well and safely the study drugs sasanlimab, palbociclib, and axitinib work for treatment of participants with advanced clear cell renal cell carcinoma (ccRCC) or translocation renal cell carcinoma (tRCC).

The name of the study drugs involved in this research study is:

* Sasanlimab (a type of monoclonal antibody)
* Palbociclib (a type of kinase inhibitor)
* Axitinib (a type of Vascular endothelial growth factor inhibitor)

DETAILED DESCRIPTION:
This single arm, Phase 2 study is to evaluate how well and safely the study drugs sasanlimab, palbociclib, and axitinib work for treatment of participants with advanced clear cell renal cell carcinoma (ccRCC) or translocation renal cell carcinoma (tRCC).

The U.S. Food and Drug Administration (FDA) has not approved sasanlimab or palbociclib as a treatment option for ccRCC or tRCC.

The U.S. FDA has approved axitinib as a treatment option for ccRCC.

The U.S. FDA has not approved the combination of sasanlimab, axitinib, and palbociclib for ccRCC or tRCC.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, urine tests, imaging scans, and electrocardiograms (ECGs).

It is expected that about 25 people will take part in this research study.

Pfizer, is supporting this research study by providing funding and the study drugs, sasanlimab, palbociclib, and axitinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable advanced or metastatic renal cell carcinoma with a clear cell component or translocation renal cell carcinoma. Patients with clear cell carcinoma and sarcomatoid histology are eligible.

  * a. For tRCC please refer to the following for eligibility definitions:

    * i. TFE3 (Xp11.2) translocation RCC: confirmed by IHC; however, FISH should be utilized if IHC is not optimal (ie, conclusive) or unavailable.
    * ii. TFEB rearranged RCC: confirmed by FISH; TFEB amplified tumors are excluded.
  * b. A formalin-fixed, paraffin-embedded (FFPE) tumor tissue block from a de novo tumor biopsy obtained during screening will be required (biopsied tumor lesion should not be a RECIST target lesion). Alternatively, a recently obtained archival FFPE tumor tissue block (not cut slides from a primary or metastatic tumor resection or biopsy) can be provided if the following criteria are met:

    * i. The biopsy or resection was performed within 1 year of registration AND
    * ii. The patient has not received any intervening systemic anti-cancer treatment from the time the tissue was obtained and registration onto the current study. If an FFPE tissue block cannot be provided as per documented regulations then 15 unstained slides (10 minimum) will be acceptable
  * c. Availability of an archival FFPE tumor tissue block from primary diagnosis specimen (if available and not provided per above). If an FFPE tissue block cannot be provided as per documented regulations, then 15 unstained slides (10 minimum) will be acceptable.
* Measurable disease as per RECIST 1.1. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Normal organ and marrow function as defined below:

  * a. Absolute neutrophil count ≥1.5×109/L
  * b. Platelets ≥100×109/L
  * c. Hemoglobin ≥9g/dL (RBC transfusions allowed)
  * d. Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) with the following exception: patients with known Gilbert disease should have a total serum bilirubin ≤ 3 x ULN
  * e. AST(SGOT)/ALT(SGPT) ≤1.5 × ULN
  * f. Creatinine clearance ≥30 mL/min according to the CKD-EPI equation. (APPENDIX C)
  * g. Urine protein <1+ by urinalysis; If ≥1+ protein or otherwise suggestive of any proteinuria above a trace amount (per local institutional standards), a random urine protein and creatinine ratio (UPCR) should be collected. A 24-hour urine collection can also be utilized for direct measurement. When multiple modalities are used, the 24-hour urine measurement takes precedence over the random UPCR; refer to section 6.2 for further guidance.
* Women of child-bearing potential and men must agree to use adequate contraception (intrauterine device or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. A negative pregnancy serum test should be obtained within 7 days of therapy initiation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation. Participants treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of sasanlimab, axitinib and palbociclib administration.
* Ability to swallow oral medications.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Treatment with the following prior therapies:

  * a. Prior systemic therapy for advanced or metastatic RCC.
  * b. Prior adjuvant or neoadjuvant therapy for RCC if disease progression or relapse has occurred within 12 months of last dose of such therapy. Treatment with an immune checkpoint inhibitor in the adjuvant setting is allowed providing more than 12 months have elapsed since last dose or completion of therapy.
  * c. Prior treatment with any immunotherapeutic agent (IL-2, IFN-α, anti-PD(L)-1, anti-CTLA-4, or any other antibody or drug targeting T-cell co-stimulation or immune checkpoint pathways).
  * d. Prior therapy with axitinib or other therapies targeting VEGF pathway in the metastatic setting (adjuvant therapy is allowed).

    e. Prior therapy with any CDK4/6 inhibitor.
* Participants with untreated brain metastases. Participants with metastatic CNS tumors may participate in this trial, if the participant is ≥ 4 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy >10 mg/day prednisone equivalents. A repeat MRI or CT brain to show stability is required.
* Wide field radiation therapy ≤ 2 weeks prior to treatment start. Prior palliative radiotherapy to metastatic non-target lesion(s) is permitted if completed at least 48hrs prior to patient registration.
* Untreated deep vein thrombosis or pulmonary embolism, or event of deep vein thrombosis or pulmonary embolism within 2 weeks of treatment start. Patient should be on at least 1 week of anticoagulation before C1D1.
* Major surgery/surgical procedures within the past 4 weeks prior to registration.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease - also see 3.2.22, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Current or prior use of immunosuppressive medication within 7 days prior to registration, except the following:

  * a. Intranasal, inhaled, topical steroids, or local steroid injections (eg. intra-articular injection).
  * b. Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent.
  * c. Steroids as premedication for hypersensitivity reactions (eg. CT scan premedication).
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3) or any history of anaphylaxis.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroidism not requiring immunosuppressive treatment are eligible.
* Vaccination within 4 weeks of the first dose of sasanlimab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza or shingles vaccines). Note, the COVID19 vaccine is not a live vaccine and permitted.
* Grade ≥3 hemorrhage within 4 weeks of registration.
* Patient with active systemic bacterial infection (requiring IV antibiotics at the time of initiating study treatment), fungal infection, or detectable viral infection. Patients with known viral infection (such as HIV) are excluded given the potential for interactions between antiretroviral agents and palbociclib and axitinib, and the potential for increased risk of life-threatening infection with therapy that is myelosuppressive. If patients are not known to have HIV, a HIV test is required prior to registration.
* Patients with known Hepatitis B or Hepatitis C infection are excluded only if there is evidence of active infection (detectable Hepatitis B surface antigen, detectable HBV DNA, or detectable Hepatitis C RNA).
* Prior allogenic or autologous stem cell or any solid organ transplant.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Participants who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant. Therapeutic use of low molecular weight heparin and factor Xa inhibitors (eg. apixaban, rivaroxaban) is permitted.
* Other malignancy diagnosed within 2 years of treatment start unless negligible risk of metastases or death according to the investigator (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma, or other malignancy not deemed to impact patients 5-year life expectancy).
* Has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), myocarditis, sudden cardiac arrest.
* Has had any major cardiovascular event within 6 months prior to treatment start, including but not limited to: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic event or New York Heart Association Class III or IV heart failure.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2 or history of long QTC syndrome. Any history of myocarditis.
* History of interstitial lung disease or other restrictive lung disease, as well as history of symptomatic respiratory condition considered clinically significant by the investigator. Individuals with a history of radiotherapy to the thorax and any history of pneumonitis will be excluded.
* Current or past tobacco users with a history of cigarette smoking greater than 30 pack-yrs (i.e., # of packs of cigarettes smoked per day × # of years patient has smoked > 30).
* Participants with a known hypersensitivity to the study compounds or to its excipients.
* Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors, including their administration within 7 days prior to treatment start (eg. Grapefruit juice or grapefruit/grapefruit-related citrus fruits [eg. Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, , clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
* Current use or anticipated need for drugs that are known strong CYP3A4/5 inducers, including their administration within 14 days prior to treatment start (eg. Phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, 23albociclib, clevidipine, St John's wort).
* Participants who have taken herbal medications within 7 days prior to treatment start. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
* Females that are pregnant or breastfeeding.
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Disease assessment will be performed every 8 weeks for the first 16 weeks, then every 12 weeks on treatment for up to 14 months
  ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.

SECONDARY OUTCOMES:
Grade 3 or Higher Treatment-Related Adverse Event (AE) Rate | AEs will be collected during study treatment, and participants will be followed for 90 days post last treatment administration, or until initiation of new cancer-directed treatment, up to 17 months.
  The percentage of participants who experienced a grade 3 or higher treatment-related AE based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms. Treatment-related AEs are defined as those rated 'Possibly", "Probably", or "Definitely" related to any of the study drugs.
Complete Response Rate (CRR) | Disease assessment will be performed every 8 weeks for the first 16 weeks, then every 12 weeks on treatment for up to 14 months
  CRR is defined as the percentage of participants achieving complete response (CR) based on RECIST 1.1 criteria. Per RECIST 1.1, CR is defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and absence of new lesions.
Deep Partial Response Rate | Disease assessment will be performed every 8 weeks for the first 16 weeks, then every 12 weeks on treatment for up to 14 months
  Deep partial response rate is defined as the percentage of participants achieving deep partial response based on RECIST 1.1. Deep partial response is defined as ≥80% reduction in target lesions by central review.
Median Progression-Free Survival (PFS) | Disease assessment will be performed every 8 weeks for the first 16 weeks, then every 12 weeks on treatment for up to 14 months
  PFS based on Kaplan-Meier method is defined as the time from protocol treatment initiation to the earlier of progression or death due to any cause. Participants alive without PD are censored at date of last disease evaluation. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Median Overall Survival (OS) | Participants will be followed for survival every 6 months after treatment discontinuation, until death or for up to 2 years, whichever comes first. Treatment duration is up to 14 months
  OS based on the Kaplan-Meier method is defined as the time from protocol treatment initiation to death due to any cause, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Berg, DO, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu